CLINICAL TRIAL: NCT06016153
Title: The Investigation of the Efficacy of Basic Life Support Education Among High School Students
Brief Title: The Efficacy of Basic Life Support Education Among Teenagers
Acronym: BLSGimiHun
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SUVM_BLS_1
Record Dates: First submitted 2023-08-17; First posted 2023-08-29 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-08

CONDITIONS: Cardiopulmonary Resuscitation; Basic Life Support; Premedical Education; Study Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instructor feedback (Active Comparator): BLS training participants will receive feedback from an experienced instructor certified by European Resuscitation Council on the depth and frequency of chest compressions, duty cycle, chest recoil and the quality of ventilation.
  Interventions: Other: Instructor feedback
- Software feedback (Experimental): BLS training participants will receive feedback based on a software (InnoMed CardioAid-1 Trainer AED, Innomed Inc., Budapest, Hungary) on the quality of chest compression (exact frequency, depth of chest compression, chest recoil and duty cycle) and tidal volume during ventilation.
  Interventions: Other: Software based feedback

INTERVENTIONS:
Other: Software based feedback — Feedback is given by the data of a software (InnoMed CardioAid-1 Trainer AED, Innomed Inc., Budapest, Hungary).
  Arms: Software feedback
Other: Instructor feedback — Feedback is given by the opinion and observation of an experienced instructor.
  Arms: Instructor feedback

SUMMARY:
Basic life support (BLS) skills are crucial not only for healthcare workers but for all lay people as well. Timely recognition of out-of-hospital cardiac arrest and the initiation of BLS by bystanders before the arrival of healthcare personnel can improve survival.

There are several methods of spreading BLS skills and improve BLS skill retention among lay people. One of these methods can be educating school children. The introduction of mandatory BLS education in schools was very effective in some European countries to increase the rate of bystander BLS.

The current study aims to investigate the efficacy of a BLS training and BLS curriculum among high school children in Hungary. Moreover, the investigators would like to optimise factors influencing skill retention in this first responder group and aim to compare two types of teaching methods: feedback given by the instructor or software-based feedback on the efficacy of chest compressions during the course.

ELIGIBILITY:
Inclusion Criteria:

* High school teenagers participating in the education of Óbudai High School, Budapest
* Written informed consent received from participants and their parents to participate in the study

Exclusion Criteria:

* No written informed consent provided by the student or parent
* Any injury or health issue influencing the efficacy of BLS skill

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
End of training BLS skill assessment based on a checklist | up to two hours
  BLS skills measured right after the training based on a checklist including the most important steps of BLS and quality of chest compression. The assessment will be performed by two instructors and the software of InnoMed CardioAid-1 Trainer AED, Innomed Inc., Budapest, Hungary.

SECONDARY OUTCOMES:
BLS skill assessment after 2 months based on a checklist | 2 months
  BLS skills measured 2 months after the training based on a checklist including the most important steps of BLS and quality of chest compression. The assessment will be performed by two instructors and the software of InnoMed CardioAid-1 Trainer AED, Innomed Inc., Budapest, Hungary.
BLS skill assessment after 6 months based on a checklist | 6 months
  BLS skills measured 6 months after the training based on a checklist including the most important steps of BLS and quality of chest compression. The assessment will be performed by two instructors and the software of InnoMed CardioAid-1 Trainer AED, Innomed Inc., Budapest, Hungary.

CONTACTS AND LOCATIONS:
Overall Officials: Endre Zima, PhD, Principal Investigator — Semmelweis University
Locations (1):
- Óbudai Gimnázium, Budapest, Hungary

REFERENCES:
- [Derived] Maar C, Zima E, Nagy B, Pal-Jakab A, Szvath P, Kiss B, Frituz G, Gal J, Merkely B, Kovacs E. The investigation of the efficiency of basic life support education among high school students: Protocol, design and implementation of an interventional, prospective longitudinal, individually randomised, parallel 1:1 grouped trial. Resusc Plus. 2024 Feb 28;18:100585. doi: 10.1016/j.resplu.2024.100585. eCollection 2024 Jun. PMID 38439933